CLINICAL TRIAL: NCT06544915
Title: Evaluating the Effects of a Synbiotic Versus Probiotic or Placebo on Gut Microbiota and Cardiometabolic Health: A Randomized Double-Blind Placebo Controlled Trial
Acronym: GUTRCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Responsible Party: Principal Investigator, Stephen J. Ives, Associate Professor, Skidmore College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2209-1044
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Blood Pressure, Body Composition, Immune Function
MeSH Terms: interventions — Synbiotics; Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind parallel study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Actives and placebos made by 3rd party in discreet containers inconspicuously labeled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Synbiotic (Experimental): synbiotic (Triplex (2x/day Probiotic capsules (2 billion CFU/capsule, ProBio5), 2x/day Capsules of gut supporting micronutrients; magnesium, vitamin c and citrus bioflavonoids (BioCleanse) and 2x/day Pre-biotic drink mixes (Slim Microbiome Activating), Plexus®, Scottsdale, AZ, USA)
  Interventions: Dietary Supplement: Synbiotic, Probiotic, Placebo
- Probiotic (Active Comparator): probiotic (2x/day probiotic capsules (2 billion CFU/capsules, NOW supplement), 2x/day capsules of collagen (Plexus), and 2x/day placebo drink mixes of corn-based maltodextrin (Plexus))
  Interventions: Dietary Supplement: Synbiotic, Probiotic, Placebo
- Placebo (Placebo Comparator): placebo control (4x/day collagen capsules and 2x/day placebo drink mixes (maltodextrin), Plexus)
  Interventions: Dietary Supplement: Synbiotic, Probiotic, Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic, Probiotic, Placebo — Use of dietary supplements to improve gut microbiome and cardiometabolic health

SUMMARY:
Accordingly, the purpose of this study is to evaluate the efficacy of 1) supplementation with Synbiotic (Plexus® Triplex), 2) commercially-available Probiotic, or 3) placebo control over 30 days on the gut microbiome, cardiometabolic health, body weight and body composition in healthy individuals.

DETAILED DESCRIPTION:
Specific Aim 1. Explore the changes in the gut microbiome using 16s rRNA sequencing to determine total bacterial counts, microbial diversity (alpha- and beta-diversity), short chain fatty acid (SCFA) concentration, circulating inflammatory biomarkers and mucosal immunity as a result of synbiotic vs. probiotic vs. placebo control.

Specific Aim 2. Document the functional changes in cardiometabolic health-related parameters; specifically, heart rate, heart rate variability (HRV), blood pressure (central and peripheral), vascular stiffness (augmentation index, AIx, and pulse wave velocity, PWV), body weight and composition, blood glucose and lipids as a result of synbiotic vs. probiotic vs. placebo control.

Specific Aim 3. Characterize the impact of synbiotic vs. probiotic vs. placebo control on perceptions of fullness/hunger, self-reported gastrointestinal health (questionnaire), and mood states.

Hypothesis: We hypothesize that the synbiotic will result in greater changes in total gut bacterial count, microbial diversity, SCFA, while reducing circulating markers of inflammation and increasing determinants of mucosal immunity. Second, the synbiotic will result in greater enhancement of cardiometabolic health over the probiotic or placebo control. Third, the synbiotic will maintain or improve perceptual indicators of fullness/hunger, gastrointestinal health, and mood states over probiotic alone or placebo control.

ELIGIBILITY:
Inclusion Criteria:

* To be included participants must be healthy, weight stable (± 4.4 lb for > 6 months prior), and 18 to 60 years of age. Participants will be expected to be relatively healthy without uncontrolled chronic disease (e.g. cardiovascular, metabolic, or pulmonary) and 1 or fewer positive risk factors for cardiovascular disease (e.g. high blood pressure, high cholesterol, etc.) as described by the American College of Sports Medicine/American Heart Association Criteria and presented in the table 1 below. Per College policy, participants who are visitors are required to be fully vaccinated against COVID-19, including a booster, and participants who are faculty, staff or students are required to be fully vaccinated against COVID-19 and receive a booster by January 24, 2022 or within 30 days of becoming eligible, unless a medical or religious exemption has been granted. Participants will be screened for eligibility by health history form in person baseline measurements are made (Figure 1). To ensure greater inclusion, ecological validity and representation, women will be included in this study; however, we will not control for menstrual cycle phase, but will document for possible statistical consideration.

Exclusion Criteria:

* Given the focus of the study those who are currently, or have recently used (<3 months), oral antibiotics or have diagnosed irritable bowel syndrome or gut/bowel maladies (short bowel syndrome, etc.) will be excluded. Subjects who present with 2 or more CVD risk factors (table above) or have uncontrolled/overt cardiovascular, pulmonary, or metabolic disease (Diabetes Mellitus), or recent blood donation (<8 weeks) will be excluded. Those who have cancer or are being treated for cancer will also be excluded. Women who are currently pregnant, breastfeeding, attempting to conceive, or amenorrheic (not associated with menopause or use of contraceptive medications) will also be excluded from the study. Anyone who is being treated for hypothyroid with levothyroxine will be excluded as one of the supplement ingredients, chromium polynicotinate, may interfere with this medication . Anyone with severe illness or compromised or suppressed immune system (e.g. taking immune suppressants, chronic viral infection or treatment) will be excluded. Anyone recently diagnosed (<1yr) with an eating disorder or food allergies will also be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Gut microbial diversity | Baseline, 15 days, 30 days
  alpha- and beta-diversity
Gut microbial count | Baseline, 15 days, 30 days
  Gut microbial species identification and quantification
Short Chain fatty acids | Baseline, 15 days, 30 days
  Short Chain Fatty Acid concentration

SECONDARY OUTCOMES:
Blood pressure | Baseline, 15 days, 30 days
  Brachial and estimated central blood pressure
Vascular Stiffness | Baseline, 15 days, 30 days
  Aortic vascular stiffness
Vascular reactivity | Baseline, 15 days, 30 days
  Using the near-infrared vascular occlusion test
Heart Rate Variability | Baseline, 15 days, 30 days
  Time and frequency domain HRV parameters
Dietary Analysis | Baseline, 15 days, 30 days
  Dietary analysis using the ASA24 system
Body Composition | Baseline, 15 days, 30 days
  Body mass, % body fat using Tanita RD 545
Blood Lipids | Baseline, 15 days, 30 days
  Blood lipid profile using Cholestech system
Salivary inflammation profile | Baseline, 15 days, 30 days
  Salimetrics ELISA for key inflammatory and immunity parameters (SIgA, IgG, alpha amylase, cortisol, c-reactive protein)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Ives, PhD, Principal Investigator — Skidmore College
Locations (1):
- Skidmore College, Saratoga Springs, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be made available upon successful publication of the findings.

REFERENCES:
- [Derived] Lang JM, Shostak ES, Quinn WK, Chervinskaya VD, Fioraso E, Smith E, Kotarsky CJ, DeBlauw JA, Lloyd JL, Ives SJ. Dyslipidemia Impacts Cardiometabolic Health and CVD Risk in a Relatively Young Otherwise Healthy Population. J Clin Hypertens (Greenwich). 2025 Jan;27(1):e14972. doi: 10.1111/jch.14972. PMID 39821451